CLINICAL TRIAL: NCT00001066
Title: A Randomized Comparative Study of Combined Zidovudine-Lamivudine (3TC) vs. the Better of ddI Monotherapy vs. Zidovudine Plus Ddl in Symptomatic HIV-1 Infected Children
Brief Title: A Comparison of Zidovudine Plus Lamivudine Versus ddI Used Alone or in Combination With Zidovudine in HIV-1 Infected Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 300
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-03

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Lamivudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Lamivudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Lamivudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To compare the efficacy of lamivudine (3TC) and zidovudine (AZT) in combination versus the better of didanosine (ddI) monotherapy or ddI/AZT combination, in symptomatic HIV-1 infected children who received less than 56 days of prior antiretroviral therapy. To evaluate the safety and tolerance of 3TC/AZT in this patient population. To determine other measures of diseases in response to the study regimens.

Currently, none of the potential treatments for HIV-1 infection has proven to be both nontoxic and effective in long-term use. However, previous studies in both adults and children have shown that 3TC combined with AZT reduced HIV load in blood and increased white blood cells. Additionally, 3TC has demonstrated a favorable safety profile.

DETAILED DESCRIPTION:
Currently, none of the potential treatments for HIV-1 infection has proven to be both nontoxic and effective in long-term use. However, previous studies in both adults and children have shown that 3TC combined with AZT reduced HIV load in blood and increased white blood cells. Additionally, 3TC has demonstrated a favorable safety profile.

Patients are randomized to receive oral 3TC/AZT, ddI/AZT, or ddI alone for at least 24 months. PER AMENDMENT 4/29/96: NOTE: Randomization to ZDV+ddI arm was terminated in Spring of 1996 based upon the results of ACTG 152. Patients on that arm will continue on blinded study drug and will be followed until the end of the study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* IVIG.
* Prophylaxis for opportunistic infection.
* EPO.
* G-CSF or GM-CSF.

Patients must have:

* Symptomatic HIV infection.
* Less than 56 days of prior antiretroviral therapy.
* Consent of parent or guardian.

NOTE:

* Co-enrollment on ACTG 219, ACTG 220, and certain ACTG opportunistic infection protocols is permitted.

Prior Medication:

Allowed:

* Up to 56 days of prior antiretroviral therapy.
* Prior immunomodulator therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy.
* Hypersensitivity to a nucleoside analog.
* Current grade 2 or higher amylase/lipase toxicity or grade 3 or 4 other toxicity.

PER AMENDMENT 4/29/96:

* Active opportunistic infection and/or serious bacterial infection at the time of entry.

Concurrent Medication:

Excluded:

* Any other anti-HIV therapy.
* Megestrol acetate ( Megace ).
* Probenecid.
* IV pentamidine.
* Human growth hormone ( hGH ).
* Systemic corticosteroids for more than 2 weeks.

Prior Medication:

Excluded:

* Investigational drug therapy within 14 days prior to study entry.

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 740
Dates: Primary Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: McKinney RE, Study Chair; Johnson GM, Study Chair
Locations (91):
- United States (87):
  - Univ of Alabama at Birmingham Schl of Med / Pediatrics, Birmingham, Alabama
  - Arkansas Children's Hosp, Little Rock, Arkansas
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - Univ of California / Davis, Sacramento, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Stanford Univ School of Medicine, Stanford, California
  - Children's Hosp of Denver, Denver, Colorado
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Yale Univ Med School, New Haven, Connecticut
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Ctr of South Florida, Fort Lauderdale, Florida
  - Univ of Florida, Gainesville, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Arnold Palmer Hosp for Children & Women, Orlando, Florida
  - All Children's Hosp, St. Petersburg, Florida
  - Univ of South Florida, Tampa, Florida
  - Saint Joseph's Hosp, Tampa, Florida
  - HRS Palm Beach County Public Health Unit, West Palm Beach, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - Mem Children's Hosp, Savannah, Georgia
  - Mount Sinai Hosp Med Ctr, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Minnesota Med School, Minneapolis, Minnesota
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - St Louis Children's Hosp, St Louis, Missouri
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - King's County Hosp Ctr / Pediatrics, Brooklyn, New York
  - SUNY - Brooklyn, Brooklyn, New York
  - Children's Hosp of Buffalo, Buffalo, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Beth Israel Med Ctr / Pediatrics, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Westchester Hosp, Valhalla, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of North Carolina at Chapel Hill / Duke Univ Med Ctr, Durham, North Carolina
  - Cincinnati Children's Hosp / Univ Hosp, Cincinnati, Ohio
  - Case Western Reserve Univ - Pediatric, Cleveland, Ohio
  - Columbus Children's Hosp, Columbus, Ohio
  - Children's Med Ctr, Dayton, Ohio
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Rhode Island Hosp / Brown Univ, Providence, Rhode Island
  - Med Univ of South Carolina, Charleston, South Carolina
  - Univ of South Carolina School of Med, Columbia, South Carolina
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Cook - Fort Worth Children's Med Ctr, Fort Worth, Texas
  - Hermann Hosp / Univ Texas Health Science Ctr, Houston, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Univ of Texas Health Science Ctr, San Antonio, Texas
  - Senetara Norfolk Gen Hosp, Norfolk, Virginia
  - Virginia Commonwealth Univ, Richmond, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (4):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Mayaguez Med Ctr, Mayagüez
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Combination therapies improve outlook for children with HIV disease. NIAID AIDS Agenda. 1997 Aug:10. PMID 11364606
- [Background] McKinney RE Jr. Ongoing and future trials of antiretroviral therapy in the pediatric AIDS clinical trials group (PACTG). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:173
- [Background] James JS. Major pediatric study stopped early: combination treatment better. AIDS Treat News. 1997 Jul 4;(No 274):5-6. PMID 11364462
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891
- [Background] Benjamin DK Jr, Miller WC, Benjamin DK, Ryder RW, Weber DJ, Walter E, McKinney RE. A comparison of height and weight velocity as a part of the composite endpoint in pediatric HIV. AIDS. 2003 Nov 7;17(16):2331-6. doi: 10.1097/00002030-200311070-00007. PMID 14571184